CLINICAL TRIAL: NCT04918446
Title: Technology-Assisted Prescription Opioid Safety Education (T-POSE)
Brief Title: Technology-Assisted Prescription Opioid Safety Education
Acronym: T-POSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Erin Winstanley, Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1705563584
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-06

CONDITIONS: Opioid Use
Keywords: Non-Medical Prescription Opioid Use

STUDY DESIGN:
Intervention Model Description: A small pilot study using a randomized clinical trial of T-POSE compared to usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-POSE (Experimental): Technology based brief educational intervention for hospitalized patients that will be discharged with an opioid prescription.
  Interventions: Other: T-POSE
- Usual Care (Other): Standard discharge instructions provided.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: T-POSE — Tablet based education and videos on opioid safety, use, and storage/disposal of the drug.
  Arms: T-POSE
Other: Usual Care — Printed instruction sheets on prescribed opioid.
  Arms: Usual Care

SUMMARY:
This study will develop a technology-based brief educational intervention for hospitalized patients that will be discharged with an opioid prescription. The Investigators will conduct a small randomized clinical trial of T-POSE to determine whether it improves patients: knowledge and reduces the incidence of Non-Medical Prescription Opioid Use (NMPOU).

DETAILED DESCRIPTION:
Non-medical use of prescription opioids (NMPOU) can be generally defined as not taking opioids as prescribed, which could occur unintentionally or intentionally. In 2014, 4.3 million adults in the United States (U.S.) were estimated to engage in NMPOU (Center for Behavioral Health Statistics and Quality 2014). Some patients may take a dose more frequently than prescribed because they were not receiving adequate pain relief from the prescribed dosage. While others may continue to take opioids longer than prescribed because their pain is persistent and/or they like the euphoric effects of opioids. According to a recently released Truven Health Analytics-NPR Health Poll, the majority (57%) of Americans have taken a prescription opioid and 35% of those had concerns (e.g., addiction, effectiveness, side effects) about prescription opioids. These findings suggest that while Americans are aware, some even concerned, of the potential dangers associated with prescription opioids that their utilization patterns continue to increase (Boddy 2017). Because opioids are prescribed by a physician, patients may believe that these medications are safe and they may be unaware of the risks associated with misuse and abuse of opioids. NMPOU may lead to increased risk of drug overdose, addiction, diversion and use of heroin. Many individuals with opioid use disorders initiated NMPOU before transitioning to heroin (Banerjee et al. 2016; Cerda et al. 2015) and report that their first exposure to an opioid was prescribed by a physician. This underscores the need for empirically-tested educational interventions that can potentially reduce NMPOU and diversion. Prescription opioids have an important role to play in health care and blanket policies to restrict access to prescription opioids are not appropriate, rather the hypothesis is that harm can be reduced by fundamentally changing our approach to opioid medication safety.

ELIGIBILITY:
Phase I Inclusion Criteria:

* Subject is being discharged from the hospital with a prescription opioid
* English Speaking
* Willing and able to use a tablet

Phase II Inclusion Criteria:

* Willing and able to provide informed written consent
* Subject is being discharged from the hospital with a prescription opioid
* English Speaking
* Willing and able to use a tablet

Exclusion Criteria:

* Visual or hearing impediment that would inhibit communication with the Study Pharmacist and use of the laptop
* Cognitive or mental state prohibiting informed consent
* Patient reported opioid use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of Non-Medical Use of a Prescription Opioid | Up to 90 days post intervention
  Self report of Yes or No to follow up questions about prescription opioid use. Yes= occurrence of Non-Medical Use of a Prescription Opioid.

SECONDARY OUTCOMES:
Occurrence of retention of knowledge on how to safe use of prescription opioids | Up to 90 days post intervention
  The number of times that a patient reports retention of materials presented.
Number of patients reporting patient satisfaction | Up to 90 days post intervention
  Overall number of subjects satisfied with T-POSE, as measured by a 5-point Patient Satisfaction questionnaire.
Reasons for non-medical use of prescription opioids | Up to 90 days post intervention
  Investigators recorded reasons for non-medical us of prescription opioids.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Winstanley, PhD, Principal Investigator — West Virginia University
Locations (2):
- United States (2):
  - Cabell Huntington Hospital (Marshall University), Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia